CLINICAL TRIAL: NCT00413452
Title: Open-Label Study to Assess the Safety and Immunogenicity of Etanercept SFP When Administered to Subjects Diagnosed With Rheumatoid Arthritis.
Brief Title: Etanercept SFP in RA Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060104
Record Dates: First submitted 2006-12-15; First posted 2006-12-19 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Etanercept; Enbrel; Amgen
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

ARMS (1):
- 50 mg (Experimental): 50 mg once weekly
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — 50 mg once weekly

SUMMARY:
Purpose of this study is to evaluate the immunogenicity and overall safety of etanercept SFP therapy administered once weekly for 24 weeks to subjects with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or older who have RA, as defined by the ACR criteria for classification of RA
* Naïve to etanercept therapy
* Able to self-inject investigational product or have a designee who can do so
* Ethical - Before any study-specific procedure, the appropriate written informed consent must be obtained Exclusion Criteria
* Receipt of Corticosteroids> 10 mg/day of prednisone (or its equivalent) during 14 days befor 1st dose of investigational product
* Receipt of MTX witin 30 days of 1st dose of investigational product
* Receipt of an other investigational drug within 30 days of 1st dose
* Receipt of TNF inhibitor therapy within 90 days of 1st dose
* Receipt of cyclophosphamide within 6 mo of 1st dose
* Current use of nonsteroidal anti-inflammatory drugs (NSAIDs) greather than the maximum recommended dose in the product info sheet
* Current use of insulin
* gnificant concurrent medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2006-12; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Etanercept seroreactivity response (ie, development of anti-etanercept antibodies) to etanercept (manufactured using the SFP) | 24 weeks

SECONDARY OUTCOMES:
Etanercept seroreactivity response to etanercept (manufactured using the SFP) | week 12
neutralizing antibodies to etanercept | week 12 and 24
Adverse events, serious adverse events (SAEs), serious infections and safety laboratory assessments | week 24

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_916_ENBREL_20060104.pdf
- See also: FDA-approved Drug Labeling — http://www.enbrel.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com